CLINICAL TRIAL: NCT03725605
Title: An Open Label Phase II Single Centre Study Investigating the Safety and Efficacy of LTX-315 and Adoptive T-cell Therapy in Patients With Advanced/Metastatic Soft Tissue Sarcoma (ATLAS-IT-04)
Brief Title: LTX-315 and Adoptive T-cell Therapy in Advanced Soft Tissue Sarcoma (ATLAS-IT-04)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C17-315-04 (ATLAS-IT-04)
Record Dates: First submitted 2018-10-02; First posted 2018-10-31 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2023-11

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — LTX-315

STUDY DESIGN:
Intervention Model Description: LTX-315 and TILs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LTX-315 plus TIL infusion (Experimental): LTX-315 intratumoural injection, TILs expansion and infusion.
  Interventions: Combination Product: LTX-315 and TILs

INTERVENTIONS:
Combination Product: LTX-315 and TILs — Intratumoural injection of LTX-315 and infusion of TILs

SUMMARY:
ATLAS-IT-04 is a two part, single arm study designed to determine the safety and effectiveness of LTX-315 to induce T-cell infiltration prior to TIL expansion in patients with soft tissue sarcoma. Following intratumoural injection of LTX-315 to a selected lesion, the lesion will be extracted for T-cell culture, expansion and infusion.

DETAILED DESCRIPTION:
Patients with advanced/metastatic tumours who have received at least one approved standard of care treatment will be recruited. All patients must have at least two lesions, one that can injected with LTX-315 and another that can used to assess response. In the first part of the study, LTX-315 will be administered intratumorally on 4-6 dosing days over a 2-4 week period to an index lesion which will be biopsied or removed after treatment for T-cell expansion. The second part will involve culturing and expanding T-cells for infusion of tumour infiltrating lymphocytes (TILs) following an induction regimen. The safety and efficacy of the LTX-315 and TIL treatment will be assessed. Patients will be followed up for 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Advanced/metastatic soft tissue sarcoma that is stable or has progressed on or after minimum 1 line of systemic treatment of advanced/metastatic disease
* At least 1 index lesion accessible for injection
* At least 1 measurable non-injected lesion that can be used for response willing to undergo repeat biopsy and tumour resection procedures
* Age between 18 and 75 years
* ECOG performance status of 0-1
* Meet following blood laboratory criteria: ANC >/= 1.5, Platelet count >/=75, - Haemoglobin >/=6mmol/L, AST and ALT </=2.5 x ULN, Creatinine </=1.5 ULN
* Willing to comply with the protocol requirements and follow-up
* Signed informed consent

Exclusion Criteria:

* A history of clinically significant active systemic autoimmune disease requiring anti inflammatory or immunosuppressive therapy within the last 3 months
* Other active malignancy within the previous 5 years except for carcinoma in situ of cervix, ductal r lobular carcinoma in situ of the breast
* Received an investigational drug within 4 weeks prior to receipt of study drug
* Received external radiotherapy or cytotoxic chemotherapy within 4 weeks prior to LTX-315 administration or have not recovered from AEs (to</= grade 1) Palliative radiotherapy to non target and lesions planned for LTX-315 injection within 4 weeks of LTX-315 administration is allowed
* Currently taking any agent with a known effect on the immune system. Stable doses of corticosteroids(up to 10mg prednisolone or equivalent) are permitted for at least 2 weeks prior to LTX-315 administration
* Any serious illness or medical condition such, but not limited to: uncontrolled infection or infection requiring antibiotics, uncontrolled cardiac failure, uncontrolled systemic and gastrointestinal inflammatory conditions, bone marrow dysplasia
* Known to test positive for HIV/AIDs, syphilis, human T-cell leukemia-lymphoma virus, active Epstein Barr, hepatitis B or C.
* history of cerebro- or cardio-vascular disorders and would be of particular risk of sequelae following a hypotensive episode
* If of child bearing potential, not willing to use effective form of contraception
* Breastfeeding and/or have a positive pregnancy test
* Donate sperm from start to 3 months after study treatment
* Expected to need any other anticancer treatment or immunotherapy during the treatment period
* Clinically active or unstable central nervous system metastases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nielsen M, Monberg T, Sundvold V, Albieri B, Hovgaard D, Petersen MM, Krarup-Hansen A, Met O, Camilio K, Clancy T, Stratford R, Sveinbjornsson B, Rekdal O, Junker N, Svane IM. LTX-315 and adoptive cell therapy using tumor-infiltrating lymphocytes generate tumor specific T cells in patients with metastatic soft tissue sarcoma. Oncoimmunology. 2023 Dec 7;13(1):2290900. doi: 10.1080/2162402X.2023.2290900. eCollection 2024. PMID 38125722

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LTX-315 plus TIL infusion
Started | 6
Completed | 4
Not Completed | 2
Not completed — Unsuccessful TIL expansion | 2

BASELINE CHARACTERISTICS:
Arm/Group | LTX-315 Plus TIL Infusion
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Total T-cell Level in Tumour Tissues From Baseline (Step 1, Week 1, Day 1) to End of Step 1 (Step 1, Week 3-5)
Description: The total T-cell level was measured at baseline and end of Step 1. Change from baseline was listed as absolute change. Data cannot be presented on subject-level and are therefore presented as the arithmetic mean value for the factor increase (+) or decrease (-) in number of cells/mm2 from baseline to end of Step 1.
Time Frame: 15 to 42 days
Population: For 1 subject evaluation was not possible due to complete necrosis of the injected lesion
Measure: Mean (Full Range); unit: factor change in cells/mm2
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 5
factor change in cells/mm2 | 1.9 [-0.6 to 6.9]

2. Primary Outcome: Adverse Events (AE) Related to LTX-315 or to the Combination of LTX-315 and Adoptive T-cell Therapy From Baseline (Step 1, Week 1, Day 1) to End of Treatment (EoT) (Step 2, Week 7)
Description: AEs were events occurring during or after administration of the IMP. AEs were coded using MedDRA version 21.1 and were classified by System Organ Class (SOC), Preferred Term (PT) and Lowest Level Term (LLT).
  Adverse events related to LTX-315 were events where causality to LTX-315 was marked on the adverse events page.
  Adverse events related to the combination of LTX-315 and adoptive T-cell therapy were events where both causality to LTX-315 and at least one of the other IMPs (TILs, Sendoxan®, Fludara® and Proleukin®) were marked on the adverse event page.
Time Frame: Up to 133 days
Population: AEs related to LTX-315 treatment were evaluated for the 6 subjects completing Step 1. AEs related to LTX-315 treatment in combination with adoptive T-cell therapy were evaluated for the 4 subjects completing Step 2.
Measure: Number; unit: events
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 6
events
  AEs related to LTX-315 treatment during Step 1. | 14
  AEs related to LTX-315 treatment in combination with adoptive T-cell therapy during Step 2: number analyzed (Participants) | 4
  AEs related to LTX-315 treatment in combination with adoptive T-cell therapy during Step 2 | 0

3. Secondary Outcome: Change in CD3+CD8+ T Cell Density in Non-injected Tumour Tissues From Baseline (Step 1, Week 1, Day 1) to EoT (Step 2, Week 7)
Description: The change is described as factor change in CD8+ cells/mm2.
Time Frame: Up to 133 days
Population: The change in CD3+CD8+ T-cells from baseline to end of Step 2 could only be evaluated for 1 subject.
Measure: Mean (Full Range); unit: factor change in CD8+ cells/mm2
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 1
factor change in CD8+ cells/mm2 | 3.3 [3.3 to 3.3]

4. Secondary Outcome: Total Number of CD3+CD8+ T-cells in TIL Infusion Product
Description: The composition of the TIL infusion product was evaluated for the subjects for whom it was possible to grow TILs.
Time Frame: 41 to 49 days between Step 1 and Step 2
Population: TIL infusion product was evaluated for the 4 subjects for whom it was possible to grow TILs. For 2 subjects it was not possible to meet the criteria of 4x10^7 cells as described in the IMPD.
Measure: Mean (Full Range); unit: million CD8+ T-cells
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 4
million CD8+ T-cells | 8032 [210 to 23177]

5. Secondary Outcome: % CD3+CD8+ T-cells of Total CD3+ in TIL Infusion Product
Description: The composition of the TIL infusion product was evaluated for the subjects for whom it was possible to grow TILs.
Time Frame: 41 to 49 days between Step 1 and Step 2
Population: The composition of the TIL infusion product was evaluated for the 4 subjects for whom it was possible to grow TILs. For 2 subjects it was not possible to meet the criteria of 4x10^7 cells as described in the IMPD.
Measure: Mean (Full Range); unit: %CD8+ of total CD3+ T-cells in TILs
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 4
%CD8+ of total CD3+ T-cells in TILs | 17 [1 to 52]

6. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: EoT (Step 2, Week 7) and up to 15 months after EoT.
Population: ORR was evaluated for the 4 subjects who progressed to Step 2.
Measure: Number; unit: participants
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 4
participants
  ORR at EoT (Step 2, Week 7) | 0
  ORR at up tp 15 months after EoT | 0

7. Secondary Outcome: Clinical Benefit Rate
Description: The clinical benefit rate (CBR) was defined as proportion of subjects who according to RECIST 1.1 had achieved complete response, partial response or stable disease at EoT (Step 2, Week 7) and up to 15 months after EoT.
  CBR was evaluated at Step 2, Week 7 and Week 13.
Time Frame: Up to 15 months
Population: The endpoint was evaluated for the 4 subjects who progressed to Step 2.
Measure: Number; unit: participants
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 4
participants
  CBR at EoT (Step 2, Week /) | 3
  CBR at up to 15 months after EoT (Week 13) | 1

8. Secondary Outcome: Best Overall Tumour Response Rate
Description: Best overall tumour response rate (BOR) was defined in the CSP as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started).
Time Frame: Assessed at Visit 25 (Step 2, Week 7, Day 42)
Population: Evaluated for the 4 subjects who progressed to Step 2.
Measure: Count of Participants; unit: Participants
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 4
Participants
  Stable disease | 3
  Progressive disease | 1

9. Secondary Outcome: Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Days from screening (Baseline) until date of progressive disease or up to 15 months after EoT.
Population: Endpoint evaluated for the 4 subjects who progressed to Step 2.
Measure: Mean (Full Range); unit: days
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 4
days | 153 [72 to 208]

10. Other Pre Specified Outcome: Number of Participants With Tumour-antigen Specific T-cells in Tumour Tissue and Peripheral Blood Mononuclear Cells
Description: Tumour-antigen Specific T-cells in Tumour Tissue and Peripheral Blood Mononuclear Cells antigen specificity assessed by enzyme-linked immuno-spot assay (ELISPOT) and flowcytometry analysis of cytokines including interferon gamma (IFNγ) and tumour necrosis factor alpha (TNF⍺)
Time Frame: Up to 15 months
Population: Endpoint evaluated for the 4 subjects who progressed to Step 2.
Measure: Number; unit: participants
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 4
participants
  Induced T-cell response against cancer testis antigens | 3
  Induced T-cell response against predicted neo-peptides | 1
  Induced T-cell response against autologous tumour cell line | 3

11. Other Pre Specified Outcome: Changes in Immunological Parameters From Baseline (Step 1, Week 1, Day 1) to 15 Months After EoT
Description: Systemic immune effect of the treatment was assessed by sequencing the TCR repertoire in the peripheral blood mononuclear cells (PBMCs), the TIL product and the biopsies. The outcome of this endpoint is described as the number of subjects for whom a systemic immune effect (in terms of expansion of a significant number of T-cell clones in the blood) was observed.
Time Frame: Up to 15 months
Population: This endpoint was evaluated for 2 subjects only.
Measure: Number; unit: participants
Arm/Group | LTX-315 plus TIL infusion
Number analyzed (Participants) | 2
participants | 2

ADVERSE EVENTS:
Time Frame: AEs were collected from the day the subject signed the informed consent and for up to 15 months.
Arm/Group | LTX-315 plus TIL infusion
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LTX-315 plus TIL infusion (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Fascial rupture (Injury, poisoning and procedural complications) | 1 (1)
Hypoglycaemia (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LTX-315 plus TIL infusion (N=6)
Anaemia (Blood and lymphatic system disorders) | 4 (8)
Neutropenia (Blood and lymphatic system disorders) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Gastric disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 3 (3)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Injection site erythema (General disorders) | 1 (1)
Injection site pain (General disorders) | 4 (9)
Localised oedema (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (6)
Oral fungal infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Blood alkaline phosphatase decreased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (2)
Blood magnesium decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 3 (3)
Transaminases decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI has the right to publish the study results in scientific or other journals, or to present the study results at professional conferences or other meetings. The PI may use the study results solely for internal research and/or educational purposes and shall not externally publish or present any such results until the earlier of (i) the date of the first study results publication, agreed by the parties and (ii) the end of the 18 month period following the completion of the study.

DOCUMENTS (2):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT03725605/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03725605/SAP_001.pdf